CLINICAL TRIAL: NCT02150941
Title: Does the BioVac Direct Suction Device Increase Identification of the Bleeding Source in Upper Gastrointestinal Bleeding: a Randomized Clinical Trial
Brief Title: Effectiveness Study of the BioVac Direct Suction Device in Upper Gastrointestinal Bleeding
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment too slow to complete the trial in a reasonable amount of time.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Michael Sai Lai Sey, MD, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 105394
Record Dates: First submitted 2014-05-22; First posted 2014-05-30 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Gastrointestinal Hemorrhage
Keywords: Upper gastrointestinal tract; Endoscopy; Endoscopic Hemostasis
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BioVac Direct Suction Device (Experimental): Experimental arm
  Interventions: Device: BioVac Direct Suction Device
- Standard Endoscopy Suction (Active Comparator): Control arm
  Interventions: Device: Standard Endoscopy Suction

INTERVENTIONS:
Device: BioVac Direct Suction Device — The BioVac Direct Suction Device (US Endoscopy) is an endoscopic device that enhances the suction power of the gastroscope.
  Arms: BioVac Direct Suction Device
Device: Standard Endoscopy Suction — Standard Endoscopy Suction refers to the suction provided on the gastroscope (Olympus EVIS EXERA III).
  Arms: Standard Endoscopy Suction

SUMMARY:
Upper endoscopy is performed for upper gastrointestinal bleeding (bleeding in the esophagus, stomach, or part of the duodenum) to identify and potentially treat the cause of bleeding. However, blood clots often make visualization difficult during endoscopy. The current practice is to try to wash off and suction up these blood clots with the endoscope. However, this is often not successful due to blood clots blocking the suction channel.

A new device has been approved by Health Canada that attaches to the endoscope and helps prevent blockage. It is believed that this device will help doctors suck out blood clots and potentially improve visualization, identification of the cause of bleeding, and possibly health outcomes, although this has never been proven. The purpose of the this clinical trial is to test whether the device works and whether it can help patients with this type of bleeding.

DETAILED DESCRIPTION:
STUDY DESIGN:

This is a randomized double blind clinical trial of the BioVac suction device versus standard endoscopy suction for UGIB. The study will be performed at London Health Sciences Center Victoria Campus and University Campus with an anticipated recruitment period of 2.5 years.

STUDY POPULATION:

All patients over the age of 18 admitted to hospital with a diagnosis of UGIB will be considered for recruitment. Patients already admitted to hospital with another diagnosis who develop UGIB will also be included.

INTERVENTION:

Patients will undergo EGD for UGIB as per standard clinical practice. If the bleeding source is not found within the first 5 minutes (timer starts once EGD passes upper esophageal sphincter) due to blood clots, the patient may benefit from additional suctioning. The patient will be randomized in blocks of 2-6 stratified by site to either the BioVac device or endoscopy suction. Those randomized to the BioVac device will use it to irrigate and suction as much blood as possible until the bleeding source is found or until the endoscopist feels that additional time would not help. Those randomized to endoscopy suction will do the same without the BioVac device. Due to the suctioning power of the study device, a placebo is not possible. Our original intention was to record the endoscopy video to blindly assess the outcome. Unfortunately, this ended up not being possible for technical reasons.

ELIGIBILITY:
Inclusion Criteria

1. Patients presenting with fresh blood hematemesis, coffee ground emesis, or melena
2. Patients with hematochezia and hypotension (systolic blood pressure < 90 mm Hg) or tachycardia (heart rate > 110 beats per minute)

Exclusion Criteria

1. Identification of a bleeding source within the first 5 minutes of the upper endoscopy or no blood seen in the upper GI tract as these patients do not require additional suctioning.
2. Age < 18.
3. No endoscopy was performed.
4. Endoscopy previously performed for current episode of UGIB.
5. Patients unable to consent and who do not have a substitute decision maker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Identification of cause of bleeding on upper endoscopy | Once at the time of endoscopy
  The cause of bleeding will be classified by location (esophagus, stomach, duodenum) and etiology (inflammation, ulcer, mass, varices, angioectasia, Dieulafoy, other).

SECONDARY OUTCOMES:
Application of any endoscopic therapy | Once at the time of endoscopy
  Treated as a dichotomous outcome (yes, no). Endoscopic therapy include injection, electrocautery, hemostatic clip, variceal banding, or Hemospray
Rebleeding | Measured once 7 days after endoscopy
  Rebleeding is defined to have occurred for any of the following: vomiting of fresh blood, shock (systolic blood pressure < 90 mm Hg or heart rate > 110 beats per minute) with melena after stabilization, or a drop in hemoglobin of > 20 g/L within 24 hours after a transfusion to a level > 70 g/L
Transfusion requirement | Measured once 7 days after endoscopy
  Total number of units of blood transfused 7 days after endoscopy
Length of hospital stay | Measured once 30 days after endoscopy
Need for interventional radiology or surgery | Measured once 30 days after endoscopy
30 day mortality | Measured once 30 days after endoscopy
Need for repeat EGD within 72 hours | Measured once 7 days after endoscopy
Procedure duration | Once at the time of endoscopy video review

OTHER OUTCOMES:
Procedure related adverse events | Measured once 48 hours after endoscopy
  Adverse events related to the EGD will be noted, including intraprocedural hypotension, oxygen desaturation, aspiration, and perforation.

CONTACTS AND LOCATIONS:
Overall Officials: Michael SL Sey, MD, Principal Investigator — London Health Sciences Centre-Victoria Campus, Western University
Locations (1):
- London Health Sciences Center, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided